CLINICAL TRIAL: NCT00310583
Title: Effects of Pregabalin on Mechanical Hyperalgesia - EPOM
Brief Title: Effects of Pregabalin on Mechanical Hyperalgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professional Associations Clinic Bergmannsheil (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-000411-10; BfArM61-3910-4030984; 4478944789; EV2005-2509
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2006-04

CONDITIONS: Tactile Hyperalgesia; Neuropathic Pain
Keywords: tactile hyperalgesia; neuropathic pain; enriched design; peripheral nerve lesion; plexus lesion; radicular lesion; spinal lesion; polyneuropathy; postzosteric neuralgia
MeSH Terms: conditions — Hyperalgesia; Neuralgia; Polyneuropathies | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The aim of this randomized placebo-controlled study is to evaluate the effects of analgetics for neuropathic pain on mechanical hyperalgesia as a kind of evoked pain. Therefore the number of responders and non-responders on pregabalin will be evaluated in respect of mechanical hyperalgesia (stimulus-response-function (SRF) on static punctual stimuli evoking pain determined via pinprick). The hypothesis is that in the placebo group the amount of non-responders is increased.

DETAILED DESCRIPTION:
This randomized controlled trial is intended to be the first in a series of trials that will assess the efficacy of drugs, which relieve neuropathic pain, on stimulus-evoked pain (here: mechanical hyperalgesia to static punctate stimuli). Most drugs in this class (e.g. Gabapentin or NMDA receptor inhibitors) have NNT beyond 3 in patients with chronic pain, due to a response rate of 30 to 50 %. One potential reason for this low overall efficacy might be the presence of different pathophysiological mechanisms in subgroups of patients, who suffer from the same disease (e.g. postherpetic neuralgia, diabetic neuropathy). These mechanisms may include central sensitization on one hand and peripheral degeneration of afferent fibers on the other hand.

In this trial, we will use a battery of mechanical and thermal Quantitative Sensory Tests (QST), using non-nociceptive and low-intensity painful stimuli, to identify a subgroup of patients with mechanical hyperalgesia. To overcome the well-known low response rate in trials with neuropathic pain patients, an enriched design comparing active drugs with placebo will be performed, including only patients with high intensity of on-going pain in combination with mechanical hyperalgesia as sequelae of different, but well defined neurological disorders. The blinded phase of the trial will be restricted to so-called responders, i.e. patients with a clinically meaningful pain reduction of at least 30% in the primary end point (mechanical hyperalgesia). The second objective of this trial is to evaluate, whether the anti-hyperalgesic effect of the active drug is dependent on the QST profile.

ELIGIBILITY:
Inclusion Criteria:

Recruitment:

* Age above 18 years;
* Neuropathic pain of at least 4/10 for at least 6 months;
* Mechanical hyperalgesia;
* One of the following diagnoses: peripheral nerve lesion, plexus lesion, radicular lesion, spinal lesion, polyneuropathy, postzosteric neuralgia;
* No nerve block or other interventional treatment for at least 4 weeks;
* Constant medication for at least 4 weeks;
* Signed informed consent;
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication;
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized.

Enrolment open titration:

* All principal inclusion criteria at recruitment
* Relevant mechanical hyperalgesia: SRF affected/control at least 2.0 with a minimal SRF of 0.8.

Enrolment double-blind phase:

* At least 30% reduction in mechanical hyperalgesia (SRF) in the open titration;
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication;
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study (see above recruitment).

Exclusion Criteria:

* Anaphylaxis on the active component or any other component of Lyrica or the placebo (Lyrica®: pregabalin, lactose-monohydrate, corn starch, talcum; capsule shells: gelatine, titanium dioxide (E 171), natriumdodecylsulfat, high dispersive siliciumdioxide, purified water; ink: shellac, black iron(II,III)-oxide (E 172), propyleneglycol, kaliumhydroxide; additionally in placebo: microcrystalline cellulose, sucrose octaacetate, magnesium stearate)
* Intake of gabapentin or pregabalin within the last 4 weeks prior to recruitment
* Any surgery within the last two months or any scheduled surgery within the study period (20 weeks);
* Concurrent unstable disease involving any system, e.g. advanced carcinoma, acute myocardial infarction, renal failure, or any other condition that in the opinion of the Investigator would deem the patient unsuitable for the study;
* History of cerebral vascular or other cerebral disease;
* Concurrent chronic or acute pain of other origin (osteoarthritis), which is not treated effectively
* Concurrent severe mental deficit, e.g. psychiatric disorders as defined by DSM IV including schizophrenia, mood disorders, organic brain syndrome, psychotic/delusional disorders, serious psychosis;
* Concurrent serious neurological disease, e.g. dementia, multiple sclerosis, or any other disease that would have impact on the ability of the patient to give their consent for the participation in the study or influences the pain perception;
* Concurrent atrioventricular block second degree or higher
* Concurrent renal failure (CLcr < 30 ml/min)
* Concurrent hereditary galactose-intolerance
* Concurrent lapp-lactase insufficiency
* Concurrent glucose-galactose-malabsorption
* Concurrent sub-optimal stabilized Diabetes Mellitus (Hb1Ac > 12%)
* Clinical apparent overdosage of opioids or psychopharmaca
* Recent history (6 months) or current evidence of alcohol or drug abuse;
* Participation in any other investigational drug or therapy study within the previous 90 days;
* Women who are pregnant or breastfeeding;
* Women with a positive pregnancy test on enrollment or prior to study drug administration;
* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study. Women practicing abstinence should use a reliable method of contraception (except birth control pills) if they choose to become sexually active during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-07; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
number of responders and non-responders in respect of mechanical hyperalgesia (stimulus-response-function (SRF) on static punctual stimuli evoking pain determined via pinprick)

SECONDARY OUTCOMES:
Degree of mechanical hyperalgesia
Ongoing pain (numerical rating scale)
Neuropathic Pain Symptom Inventory score
Additional QST (qualitative sensory testing) variable CDT = cold detection threshold,
Additional QST (qualitative sensory testing) variable HDT = heat detection threshold
Additional QST (qualitative sensory testing) variable TSL = thermal sensory limen
Additional QST (qualitative sensory testing) variable PHS = number of paradoxical heat sensations during the TSL Procedure
Additional QST (qualitative sensory testing) variable CPT = cold pain threshold
Additional QST (qualitative sensory testing) variable HPT = heat pain threshold
Additional QST (qualitative sensory testing) variable MDT = mechanical detection threshold
Additional QST (qualitative sensory testing) variable MPT = mechanical pain threshold
Additional QST (qualitative sensory testing) variable ALL = dynamic mechanical allodynia
Additional QST (qualitative sensory testing) variable WUR = windup ratio
Additional QST (qualitative sensory testing) variable VDT = vibration detection threshold
Additional QST (qualitative sensory testing) variable PPT = pressure pain threshold)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. MD., Study Director — Professional Associations Clinic Bergmannsheil , Dept. of Pain Therapy
Locations (17):
- Germany (17):
  - Berufsgenossenschaftliche Kliniken Bergmannsheil, Dept. of Anaesthesiology, Intensive Care and Pain Therapy, Dept. of Pain Therapy, Bochum
  - Pain Therapy, Dept. of Anaesthesiology and Intensive Care Medicine, University of Cologne, Cologne
  - University Hospital of Duesseldorf, Dept. of Paintherapy, Dept. of Anaesthesiology, Düsseldorf
  - Dept. of Anaesthesiology, University Hospital of Erlangen, Erlangen
  - Insitute of Physiology and Experimental Pathophysiology, Erlangen
  - Neurological University Hospital, University of Freiburg, Freiburg im Breisgau
  - Dept. of Neuroradiology, Neurological Health Care Center, University Hospital of Heidelberg, Heidelberg
  - Dept. of Neurology, Neurological Section, Pain Research and Therapy, Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Health Care Centre, Dept. of Neurology, Johannes Gutenberg University of Mainz, Mainz
  - DRK - Pain Centre Mainz, Mainz
  - Pain Therapy, Dept. of Anaestesiology and Intensive Care Medicine, Clinical Medicine Mannheim, University of Heidelberg, Mannheim
  - Interdisciplinary Dept. of Pain Management, Dept. of Anaesthesiology, Ludwig-Maximilians-University, Munich
  - Dept. of Neurology, Universtity Hospital TU Munich, Munich
  - Anesthesiology and Surgical Intensive Care Medicine, University of Muenster, Münster
  - Dept. of Anaesthesia and Transfusion Medicine, University of Tuebingen, Tübingen
  - Dept. of Neurology, University of Ulm, Ulm
  - Neurological Hospital, University of Wuerzburg, Würzburg

REFERENCES:
- See also: German Ministry of Education and Research — http://www.bmbf.de/
- See also: German Federal Institute for Drugs and Medical Devices — http://www.bfarm.de
- See also: Ethics Committee, Medical Department of the Ruhr-University Bochum — http://www.ruhr-uni-bochum.de/ethik/